CLINICAL TRIAL: NCT02454140
Title: Phase I Trial of Adaptive Stereotactic Body Radiotherapy (SBRT) Dose Escalation in Pancreatic Cancer
Brief Title: Stereotactic Body Radiotherapy Dose Escalation in Pancreatic Cancer
Acronym: SBRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, James D. Murphy, MD, MS, Associate Clinical Professor, Radiation Medicine, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 140103
Record Dates: First submitted 2015-01-11; First posted 2015-05-27 (Estimated); Results first posted 2025-09-12 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-08

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Cohort 1 (Experimental): SBRT 40 Gy in 5 fractions
  Interventions: Radiation: SBRT
- Cohort 2 (Experimental): SBRT 45 Gy in 5 fractions (starting dose level)
  Interventions: Radiation: SBRT
- Cohort 3 (Experimental): SBRT 50 Gy in 5 fractions
  Interventions: Radiation: SBRT
- Cohort 4 (Experimental): SBRT 55 Gy in 5 fractions
  Interventions: Radiation: SBRT
- Cohort 5 (Experimental): SBRT 60 Gy in 5 fractions
  Interventions: Radiation: SBRT

INTERVENTIONS:
Radiation: SBRT — Fixed five-fraction stereotactic radiotherapy

SUMMARY:
This study is to determine the maximum tolerated dose (MTD) of five fraction stereotactic radiotherapy (SBRT) in pancreatic cancer.

DETAILED DESCRIPTION:
This trial is designed to find the maximum tolerated dose of radiation under a fixed 5-fraction SBRT regimen escalating the dose from 40 Gy in 5 fractions, to 60 Gy in 5 fractions, at 5 Gy intervals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis: Histologically-proven invasive adenocarcinoma of the pancreas.
* Disease Status: Medically unresectable (any stage), or locally advanced (stage III).
* Tumor Location: Primary tumor may be located anywhere in the pancreas.
* Treatment eligibility: The patient must be able to have fiducial markers implanted into the pancreatic tumor, and receive radiation regimen as specified in the protocol.
* Performance Level: Karnofsky Performance Status ≥ 60
* Adequate Renal Function Defined As: Serum creatinine ≤ 1.5 x upper limit of normal
* Informed Consent: All subjects must sign a written informed consent.

Exclusion Criteria:

* Pregnancy or Breast-Feeding: Pregnant or breast-feeding women will not be entered on this study due to risks of fetal and teratogenic adverse events. (Note: Serum Pregnancy tests must be obtained in women of child bearing potential). Sexually active females may not participate unless they have agreed to use an effective contraceptive method (such as abstinence, diaphragm, condom, or intrauterine device) to prevent pregnancy for the duration of the study.
* Life expectancy < 6 months
* The patient cannot have had prior radiation therapy to the thorax or upper abdomen.
* Incarcerated individuals
* Subjects unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-06-20 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Murphy, MD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD Moores Cancer Center, La Jolla, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
Started | 3 | 16 | 11 | 0 | 0
Completed | 3 | 16 | 11 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: This dose-escalation study only enrolled patients in the first three cohorts.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5 | Total
Number analyzed (Participants) | 3 | 16 | 11 | 0 | 0 | 30
Age, Continuous [Mean (Full Range); unit: years] | 71.3 [53 to 82] | 70.3 [42 to 90] | 77.2 [62 to 89] |  |  | 72.9 [42 to 90]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 5 |  |  | 12
  Male | 1 | 11 | 6 |  |  | 18
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 3 | 16 | 11 |  |  | 30

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose
Description: The purpose of this study is to determine the maximum tolerated dose of five fraction stereotactic radiotherapy (SBRT) in pancreatic cancer.
Time Frame: From date of randomization to observed dose limiting toxicity (DLT) in 20% of patients assessed up to 3 years
Population: Patients we're treated at 3 dose levels (40, 45, and 50 Gy). The dose-limiting toxicity for the study was 50 Gy
Measure: Number; unit: Gray
Groups:
- All Participants: SBRT: Fixed five-fraction stereotactic radiotherapy
Arm/Group | All Participants
Number analyzed (Participants) | 30
Gray | 50

ADVERSE EVENTS:
Time Frame: 6 years
Arm/Group | Cohort 1 | Cohort 2 | Cohort 3 | Cohort 4 | Cohort 5
All-Cause Mortality (participants affected / at risk) | 3/3 | 16/16 | 11/11 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/3 | 2/16 | 0/11 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/3 | 0/16 | 0/11 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (N=3) | Cohort 2 (N=16) | Cohort 3 (N=11) | Cohort 4 (N=0) | Cohort 5 (N=0)
Upper gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 4 upper GI bleed
Hematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Grade 5 hematemesis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-22): https://cdn.clinicaltrials.gov/large-docs/40/NCT02454140/Prot_SAP_000.pdf